CLINICAL TRIAL: NCT05756166
Title: Phase I/IIa Clinical Trial Evaluating the Safety and Efficacy of Rintatolimod Combined With IFNα2b (Bioferon®) to Enhance the Effectiveness of Pembrolizumab in Patients With Metastatic Triple Negative Breast Cancer
Brief Title: Rintatolimod, Celecoxib and Interferon Alpha 2b With Pembrolizumab For the Treatment of Patients With Metastatic or Unresectable Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding ended
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-3010822; NCI-2023-01262 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3010822 (Other: Roswell Park Cancer Institute); P01CA234212 (NIH)
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Carcinoma; Unresectable Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Biopsy; Specimen Handling; Celecoxib; Interferon alpha-2; Magnetic Resonance Spectroscopy; pembrolizumab; poly(I).poly(c12,U)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort I (CKM, pembrolizumab) (Experimental): Patients receive rintatolimod IV, celecoxib PO, interferon alpha-2b IV on days 0, 1, and 2 of week 1 and days 7, 8, and 9 of week 2 on study. Patients receive pembrolizumab IV on day 9 and then every 3 weeks after that for up to 4 doses on study. Patients also undergo CT scan or MRI at screening and follow-up and undergo blood sample collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Celecoxib; Procedure: Computed Tomography; Biological: Interferon Alpha-2; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Drug: Rintatolimod
- Cohort II (CMK, early pembrolizumab) (Experimental): Patients receive rintatolimod IV, celecoxib PO, and interferon alpha-2b IV on days 0, 1, and 2 of week 1 and days 7, 8, and 9 of week 2 on study. Patients receive pembrolizumab IV on day 2 of week 1 and then every 3 weeks beginning in week 4 on study. Patients also undergo CT scan or MRI at screening and follow-up, undergo blood sample collection during screening and on study, and may undergo tumor biopsy at screening and follow-up.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Celecoxib; Procedure: Computed Tomography; Biological: Interferon Alpha-2; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Drug: Rintatolimod

INTERVENTIONS:
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
  Arms: Cohort II (CMK, early pembrolizumab)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Celecoxib — Given PO
  Other Names: Benzenesulfonamide, 4-[5-(4-methylphenyl)-3-(trifluoromethyl)-1H-pyrazol-1-yl]-; Celebrex; SC-58635; YM 177
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Biological: Interferon Alpha-2 — Given IV
  Other Names: Alpha-2-Interferon; Alpha-2a Interferon; IFN-Alpha-2; IFN-AlphaA; IFNA2; IFNA2 Protein; Interferon Alpha 2; Interferon Alpha 2a; Interferon Alpha 2b; Interferon Alpha A; Interferon Alpha-A; LeIF A
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Rintatolimod — Given IV
  Other Names: Ampligen; Atvogen

SUMMARY:
This phase I/IIa trial tests the safety, side effects, and best dose of chemokine modulation therapy (CKM) (rintatolimod, celecoxib, and interferon alpha 2b) in combination with pembrolizumab for the treatment of patients with triple negative breast cancer that has spread from where it first started (primary site) to other places in the body (metastatic) or that cannot be removed by surgery (unresectable). CKM drugs such as rintatolimod and interferon alpha 2b work to modify the immune response and tumor-related processes, including tumor cell growth, blood vessel growth, and metastasis. Celecoxib is an anti-inflammatory drug that can cause cell death and may reduce the growth of blood vessels tumors need to grow and spread. Immunotherapy such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving CKM therapy prior to pembrolizumab may direct the immune cells to the cancer cells and maximize the effectiveness of pembrolizumab in patients with metastatic or unresectable triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety profile of modified CKM (celecoxib, rintatolimod and interferon alpha-2b) regimen (replacement of INTRON [registered trademark] A, using alternative source of interferon alpha-2b [IFNalpha2b]) combined with pembrolizumab therapy in metastatic triple negative breast cancer patients.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of the CKM in combination with pembrolizumab in patients with metastatic triple negative breast cancer (mTNBC) as compared to historic outcomes of pembrolizumab and other anti-PD1/PD-L1 therapies alone, as determined by secondary measures of efficacy including:

Ia. Progression-free survival (PFS); Ib. Overall survival (OS); Ic. Overall response rate (ORR) to the combination therapy using Immune Modulated Response Evaluation Criteria in Solid Tumors (iRECIST); Id. Disease control rate (DCR) using iRECIST.

EXPLORATORY OBJECTIVES:

I. Examine the immune analysis profile of CKM and pembrolizumab combination:

Ia. Examine the relationship of infiltrating CD4+ and CD8+ T cells and other immune and genetic markers, and their associated PD-1, CD45RA or CD45RO levels; Ib. Correlate PD-L1 expression within both neoplastic and nonneoplastic stromal elements of the tumor microenvironment to PFS, OS, ORR and adverse events (AEs); Ic. Correlate immune panel results with ORR, PFS, OS and AEs.

II. Comparison of response assessment criteria for a prospective analysis:

IIa. Response evaluation criteria in solid tumors (RECIST) 1.1 response assessment; IIb. iRECIST response assessment.

OUTLINE: This is a phase I dose escalation study of interferon alpha-2b followed by a phase II study. Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients receive rintatolimod intravenously (IV), celecoxib orally (PO), interferon alpha-2b IV on days 0, 1, and 2 of week 1 and days 7, 8, and 9 of week 2 on study. Patients receive pembrolizumab IV on day 9 and then every 3 weeks after that for up to 4 doses on study. Patients also undergo computed tomography (CT) scan or magnetic resonance imaging (MRI) at screening and follow-up and undergo blood sample collection during screening and on study.

COHORT II: Patients receive rintatolimod IV, celecoxib PO, and interferon alpha-2b IV on days 0, 1, and 2 of week 1 and days 7, 8, and 9 of week 2 on study. Patients receive pembrolizumab IV on day 2 of week 1 and then every 3 weeks beginning in week 4 on study. Patients also undergo CT scan or MRI at screening and follow-up, undergo blood sample collection during screening and on study, and may undergo tumor biopsy at screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age
* Have pathologically confirmed diagnosis of PDL-1-negative or PDL1 positive unresectable or metastatic TNBC with no curative treatment options
* Have been informed of other treatment options
* Patient has lesion that can be biopsied and is willing to undergo the procedure as part of the protocol. Note: For cohort 1 and cohort 2: Patient with accessible tumor will be offered optional pre-treatment and post-treatment biopsies. Biopsies are mandatory for cohort 3
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to swallow and retain oral medication
* Have measurable disease per RECIST 1.1 criteria present
* Any line of therapy allowed, radiologically confirmed progression
* No cancer-directed therapy for at least 3 weeks prior to study treatment (bone-directed therapies are allowed)
* Platelets >= 100,000/uL
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1500/uL
* Total bilirubin =< institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X institutional ULN
* Creatinine < ULN or, creatinine clearance >= 50 mL/min per Cockcroft-Gault equation for patients with creatinine levels greater than ULN
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients currently treated with systemic immunosuppressive agents, including steroids (greater than equivalent of 10 mg daily of prednisone), are ineligible until 3 weeks after removal from immunosuppressive treatment. (Inhaled steroids are allowed.)
* Patients with active autoimmune disease or history of transplantation
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Patients with known serious mood disorders. (Major depression diagnosis is an exclusion. Other stable mood disorders on stable therapy for > 6 months or not requiring therapy may be allowed after consultation with the principal investigator.)
* Cardiac risk factors including:

  * Patients experiencing cardiac event(s) (acute coronary syndrome, myocardial infarction, or ischemia) within 3 months of signing consent. While our published clinical studies involving short-term CKM did not indicate increased risk of cardiac events, the CKM can induce flu-like symptoms, providing justification for its avoidance in patients with recent cardiac events
  * Patients with a New York Heart Association classification of III or IV
  * Patients with a history of stroke
* History of upper gastrointestinal ulceration, upper gastrointestinal bleeding, or upper gastrointestinal perforation within the past 3 years
* Prior allergic reaction or hypersensitivity to nonsteroidal antiinflammatory drug (NSAIDs) or any drugs administered on protocol
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug
* Any patients with a positive antinuclear antibodies test will be excluded from study
* Has a known history of human immunodeficiency virus (HIV) infection
* Concurrent active hepatitis B (defined as hepatitis B antigen [HBsAg] positive and/or detectable hepatitis B virus [HBV] deoxyribonucleic acid [DNA]) and hepatitis C virus (defined as anti-hepatitis C virus [HCV] antibody [Ab] positive and detectable HCV ribonucleic acid [RNA]) infection. Note: Hepatitis B and C screening tests are not required unless known history of HBV and HCV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  The dose limiting toxicities will be summarized by cohort using frequencies and relative frequencies.

SECONDARY OUTCOMES:
Progression-free survival | From the start of post-chemokine modulation (CKM) therapy therapy until disease progression, death, or lst follow-up, assessed up to 2 years
  Will be summarized using standard Kaplan-Meier methods, with estimates of the median survival obtained with 90% confidence intervals.
Overall response rate | From the start of study treatment until end of treatment or disease progression/recurrence, assessed up to 2 years
  Evaluated using Immune Modulated Response Evaluation Criteria in Solid Tumors. Will be summarized using frequencies and relative frequencies, and obtained with 90% confidence intervals.
Overall survival | From the start of post-CKM therapy until death due to any cause or last follow up, assessed up to 2 years
  Will be summarized using standard Kaplan-Meier methods, with estimates of the median survival obtained with 90% confidence intervals.
Disease control rate | Up to 2 years
  Will be summarized using frequencies and relative frequencies and obtained with 90% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Ellis Levine, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT05756166/ICF_000.pdf